CLINICAL TRIAL: NCT07064447
Title: National Prospective Registry of Direct Cholangiopancreatoscopy by Single Operator
Brief Title: Spanish Registry of Direct Cholangiopancreatoscopy by Single Operator
Status: Not yet recruiting | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Spanish Society of Digestive Endoscopy (Other)
Responsible Party: Sponsor
Other Study IDs: Pl-24-022
Record Dates: First submitted 2025-05-21; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Cholangiocarcinoma; Cholangiopathy; Biliary Stricture; Choledocholithiasis; Pancreatic Cancer
Keywords: Cholangiopancreatoscopy; indeterminate biliary stricture; choledocholitiasis; pancreatic cancer; cost-effectiveness; algorithm
MeSH Terms: conditions — Cholangiocarcinoma; Choledocholithiasis; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with biliopancreatic pathology undergoing cholangiopancreatoscopy: Patients with biliopancreatic pathology who undergo cholangiopancreatoscopy, are over 18 years of age, and have signed the informed consent
  Interventions: Procedure: Cholangiopancreatoscopy

INTERVENTIONS:
Procedure: Cholangiopancreatoscopy — Direct cholangiopancreatoscopy by single operator

SUMMARY:
Endoscopic ultrasound (EUS) and endoscopic retrograde cholangiopancreatography (ERCP) remain fundamental tools for the diagnosis and treatment of many pancreatobiliary diseases.

However, there are situations in which these procedures face limitations, such as the evaluation of indeterminate ductal strictures or the management of complex choledocholithiasis.

Direct visualization of the biliary and pancreatic ducts has proven to be a useful and effective alternative in such cases. It also has a safety profile comparable to conventional ERCP, with only a slight increase in the incidence of adverse events.

Nevertheless, due to the associated increase in costs, most centers have adopted a stepwise approach in their diagnostic and therapeutic algorithms, using this technique only after multiple ERCPs.

Although the evidence is still limited, recent studies suggest that early use of direct cholangiopancreatoscopy could be a cost-effective strategy due to its increased efficacy.

In this regard, collecting data on direct cholangiopancreatoscopy would be of interest to generate robust conclusions on cost-effectiveness in routine clinical practice.

This study aims to objectively assess the real-world use of direct cholangiopancreatoscopy in our setting, with the goal of confirming technical aspects, efficacy, and safety, and ultimately conducting cost-effectiveness evaluations to determine the optimal point in the algorithm at which this technique should be introduced.

DETAILED DESCRIPTION:
Endoscopic procedures, more specifically endoscopic ultrasound (EUS) and endoscopic retrograde cholangiopancreatography (ERCP), remain fundamental in the study and/or treatment of many pancreatic and biliary tract diseases.

However, there are certain situations in which these procedures face limitations, whether due to the characteristics of the pathology itself or the technique's constraints. This is the case, for example, in the evaluation of indeterminate ductal strictures or the management of complex choledocholithiasis, where the diagnostic or therapeutic yield is often suboptimal.

Direct visualization of the biliary and pancreatic ducts has been shown to be a useful and effective alternative in such scenarios. Its safety profile is similar to that of conventional ERCP, with only a slight increase in the incidence of adverse events.

Despite this, the increased costs associated with this technique have led most centers to adopt a stepwise approach in their clinical algorithms. In general, conventional ERCP is used initially, and direct cholangiopancreatoscopy is only considered after several failed ERCPs.

While the economic evidence remains limited, recent studies suggest that early implementation of this technique could be a cost-effective solution, due to its high efficacy and the potential reduction in the total number of procedures required.

In this context, collecting data on the use of direct cholangiopancreatoscopy would be valuable to generate robust conclusions regarding the real-world efficacy and cost-effectiveness of the technique in routine clinical practice data that is currently lacking.

This study aims to objectively assess the real-world use of direct cholangiopancreatoscopy in our setting, to confirm technical, efficacy, and safety data for both its diagnostic and therapeutic indications, and ultimately to perform cost-effectiveness analyses to help determine the optimal point within the clinical algorithm at which this technique should be introduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cholangiopancreatoscopy at the participating centers from 1 June 2025 will be included.
* Be over 18 years of age.
* Provide signed informed consent.

Exclusion Criteria:

* Age under 18 years.
* Lack of availability of signed informed consent.
* Impossibility of follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biliopancreatic pathology fo whom a cholangiopancreatoscopy is performed in hospitals in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Timing of cholangioscopy in the management of complex biliary pathologies. | Through study completion, an average of 1 year.
  To determine the optimal timing for the use of direct cholangiopancreatoscopy in the management of complex choledocholithiasis and the evaluation of indeterminate biliary strictures.

SECONDARY OUTCOMES:
Diagnostic and therapeutic success rate in cholangioscopy. | Through study completion, an average of 1 year
  To assess whether the effectiveness of the main indications for direct cholangiopancreatoscopy in our setting (complex choledocholithiasis, evaluation of indeterminate strictures) aligns with the currently available evidence.
  The evaluation will include direct visualization of target lesions, diagnostic accuracy, number and usefulness of the biopsies, diagnosis achieved and stone clearance rate.
Incidence of procedure-related adverse events following cholangioscopy. | 1 month
  To evaluate the rate of adverse events associated with direct cholangiopancreatoscopy for its main indications in our setting (complex choledocholithiasis, evaluation of indeterminate strictures) and to assess whether these findings align with the currently available evidence.
  The evaluation will include post-ERCP pancreatitis, cholangitis, bleeding, perforation, mortality.
Incremental cost-effectiveness ratio of early cholangioscopy compared to repeated ERCPs. | Through study completion, an average of 1 year.
  To compare early cholangioscopy versus repeated ERCPs in both diagnostic and therapeutic indications for complex biliary pathologies, in terms of cost-effectiveness.
  The analysis will consider procedure-related expenses (ERCPs, Cholangioscopy), hospital admissions and length of hospitalization, ICU admission, number of outpatient visits, need for surgery, imaging studies, success rate and time until complete resolution or end of management.

CONTACTS AND LOCATIONS:
Overall Officials: Eloi Nuñez-Garcia, MD, Principal Investigator — Germans Trias i Pujol Hospital

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in cholangiopancreatoscopy and biliopancreatic diseases. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
  Data requests can be submitted starting 10 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 10 months and ending 2 years after the publication of results.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.

REFERENCES:
- [Background] Alrajhi S, Barkun A, Adam V, Callichurn K, Martel M, Brewer O, Khashab MA, Forbes N, Almadi MA, Chen YI. Early cholangioscopy-assisted electrohydraulic lithotripsy in difficult biliary stones is cost-effective. Therap Adv Gastroenterol. 2021 Jul 23;14:17562848211031388. doi: 10.1177/17562848211031388. eCollection 2021. PMID 34804204
- [Background] Sljivic I, Trasolini R, Donnellan F. Cost-effective analysis of preliminary single-operator cholangioscopy for management of difficult biliary stones. Endosc Int Open. 2022 Sep 14;10(9):E1193-E1200. doi: 10.1055/a-1873-0884. eCollection 2022 Sep. PMID 36118645
- [Background] Deprez PH, Garces Duran R, Moreels T, Furneri G, Demma F, Verbeke L, Van der Merwe SW, Laleman W. The economic impact of using single-operator cholangioscopy for the treatment of difficult bile duct stones and diagnosis of indeterminate bile duct strictures. Endoscopy. 2018 Feb;50(2):109-118. doi: 10.1055/s-0043-121268. Epub 2017 Nov 24. PMID 29172216
- [Background] Wen LJ, Chen JH, Xu HJ, Yu Q, Liu K. Efficacy and Safety of Digital Single-Operator Cholangioscopy in the Diagnosis of Indeterminate Biliary Strictures by Targeted Biopsies: A Systematic Review and Meta-Analysis. Diagnostics (Basel). 2020 Sep 2;10(9):666. doi: 10.3390/diagnostics10090666. PMID 32887436
- [Background] Turowski F, Hugle U, Dormann A, Bechtler M, Jakobs R, Gottschalk U, Notzel E, Hartmann D, Lorenz A, Kolligs F, Veltzke-Schlieker W, Adler A, Becker O, Wiedenmann B, Burgel N, Troger H, Schumann M, Daum S, Siegmund B, Bojarski C. Diagnostic and therapeutic single-operator cholangiopancreatoscopy with SpyGlassDS: results of a multicenter retrospective cohort study. Surg Endosc. 2018 Sep;32(9):3981-3988. doi: 10.1007/s00464-018-6141-0. Epub 2018 Mar 12. PMID 29532224
- [Background] Korrapati P, Ciolino J, Wani S, Shah J, Watson R, Muthusamy VR, Klapman J, Komanduri S. The efficacy of peroral cholangioscopy for difficult bile duct stones and indeterminate strictures: a systematic review and meta-analysis. Endosc Int Open. 2016 Mar;4(3):E263-75. doi: 10.1055/s-0042-100194. Epub 2016 Feb 4. PMID 27004242
- [Background] Kim HJ, Choi HS, Park JH, Park DI, Cho YK, Sohn CI, Jeon WK, Kim BI, Choi SH. Factors influencing the technical difficulty of endoscopic clearance of bile duct stones. Gastrointest Endosc. 2007 Dec;66(6):1154-60. doi: 10.1016/j.gie.2007.04.033. Epub 2007 Oct 22. PMID 17945223
- [Background] Navaneethan U, Njei B, Lourdusamy V, Konjeti R, Vargo JJ, Parsi MA. Comparative effectiveness of biliary brush cytology and intraductal biopsy for detection of malignant biliary strictures: a systematic review and meta-analysis. Gastrointest Endosc. 2015 Jan;81(1):168-76. doi: 10.1016/j.gie.2014.09.017. Epub 2014 Nov 1. PMID 25440678